CLINICAL TRIAL: NCT06263309
Title: Mid-Term Radiological Outcomes of Femoral Neck Fractures Treated With Osteosynthesis: A Comparative Analysis
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Samet Gokceoglu, Principal investigator, Istanbul University
Other Study IDs: Femoralneckfracture
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Femoral Neck Fractures; Femoral Neck Shortening
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good Functional Score: Harris hip score > 80
  Interventions: Diagnostic Test: Femoral neck shortening measurement
- Bad Functional Score: Harris Hip score < 80
  Interventions: Diagnostic Test: Femoral neck shortening measurement

INTERVENTIONS:
Diagnostic Test: Femoral neck shortening measurement — We examine femoral neck shortening in patients with femoral neck fractures.

SUMMARY:
OBJECTIVES: This study assesses the efficacy of dynamic hip screw (DHS) versus cannulated screws for femoral neck fractures, focusing on femoral neck shortening, avascular necrosis (AVN) incidence, and functional outcomes.

METHODS:

Design: Retrospective cohort study. Setting: Academic Level I Trauma Center. Patient Selection Criteria: Included were patients with femoral neck fractures treated with DHS or cannulated screws, with follow-up data available.

Outcome Measures and Comparisons: Main outcomes were femoral neck shortening, incidence of AVN, and Harris Hip Score (HHS) for functional assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 80 years and younger
* Minimum of 2 years' follow-up
* Diagnosed with a femoral neck fracture
* Treated with either cannulated screws or a Dynamic Hip Screw (DHS).

Exclusion Criteria:

* Patients with multiple fractures in the same extremity
* Presence of malignancy
* Diagnosis of osteoporosis
* Systemic inflammatory or metabolic diseases
* Infection or malignancy in the hip joint
* Insufficient medical records
* Patients unwilling to participate in the study.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent osteosynthesis for femoral neck fracture (FNF)
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Harris Hip score | minimum 2 years
  Hip functional score

CONTACTS AND LOCATIONS:
Locations (1):
- University, Istanbul, Turkey (Türkiye)